CLINICAL TRIAL: NCT06005402
Title: A Phase 1a, Randomized, Double-Blind, Placebo-Controlled, Single Site, Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of CSX-1004 Injection in Healthy Adults
Brief Title: Safety, Tolerability, and Pharmacokinetics of CSX-1004
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cessation Therapeutics, Inc. (Industry)
Collaborators: Dr. Vince Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CSX-1004.101
Record Dates: First submitted 2023-08-04; First posted 2023-08-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Opioid Overdose; Opioid Use Disorder
MeSH Terms: conditions — Opiate Overdose; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Single ascending dose study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CSX-1004 (Experimental): Single doses of CSX-1004 Injection
  Interventions: Biological: CSX-1004
- Placebo (Placebo Comparator): Sterile saline for injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CSX-1004 — Recombinant human immunoglobulin G (IgG) 1λ monoclonal antibody specific for fentanyl and structurally related fentanyl analogs
  Arms: CSX-1004
Biological: Placebo — Sterile saline for injection
  Arms: Placebo

SUMMARY:
This is a Phase 1a, randomized, double-blind, single ascending dose study, designed to assess the safety, tolerability, and PK of a single CSX-1004 injection, administered by IV infusion across a range of doses in healthy adult subjects. The study will have 3 phases: Screening, Inpatient Treatment, and Outpatient Follow-up.

The primary objective of the study is to determine the safety and tolerability of CSX-1004 Injection administered by intravenous (IV) infusion across a range of doses in healthy adult subjects.

The secondary objective of the study is to determine the pharmacokinetics (PK) of CSX-1004 Injection administered by IV infusion across a range of doses in healthy adult subjects.

ELIGIBILITY:
Major Inclusion Criteria:

* Healthy male or female subjects, aged 18 to 50 years, inclusive,
* Minimum weight of 50.0 kg and maximum weight of 100.0 kg
* Body mass index (BMI) within the range of 18.0 to 32.0 kg/m2, inclusive

Major Exclusion Criteria:

* Positive UDS for substances of abuse (including alcohol) at Screening or admission to the Treatment Phase
* Current daily cigarette smoker within 3 months of Screening. Social smoking, as defined by non-daily use of nicotine-containing products, is permitted.
* History or presence of any clinically significant cardiac, psychiatric, endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, renal, or other major disease or illness at Screening, which in the opinion of the Investigator, might jeopardize the safety of the subject or the validity of the study results.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (AEs), serious AEs, and AEs leading to discontinuation | 5 months
  Incidence, intensity, and causality of adverse events
Clinical laboratory assessments | 5 months
  Hematology, biochemistry, and urinalysis
Vital signs | 5 months
  Blood pressure and pulse rate
12-Lead electrocardiogram | 5 months
  Variables will include ventricular heart rate and the PR, QRS, QT, QTcB and QTcF intervals
Physical examination | 5 months
  Complete physical examination, assessing the subject's overall health and physical condition
Infusion site examination | 6 days
  Infusion site will be visually inspected for evidence of erythema, edema, itching, pain, infection, bleeding, abnormal healing, and any other abnormalities

SECONDARY OUTCOMES:
Cmax | 4 months
  Maximum serum concentration
AUCinf | 4 months
  Area under the curve from time zero extrapolated to infinity
AUClast | 4 months
  Area under the curve from time zero to the last measurable concentration
Tmax | 4 months
  Time to maximum serum concentration
t1/2 | 4 months
  beta terminal elimination half-life

OTHER OUTCOMES:
Immunogenicity | 4 months
  Proportions of subjects who are positive (above the limits of quantitation) and negative (below the limits of quantitation) for anti-CSX-1004 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hull, MD, Principal Investigator — Dr. Vince Clinical Research
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No